CLINICAL TRIAL: NCT04699240
Title: A Prospective, Case-controlled Randomized Study of Human Reproductive Tract Active Lactobacillus in Adjuvant Treatment of Recurrent Vulvovaginal Candidiasis.
Brief Title: Study of Lactobacillus in Adjuvant Treatment of RVVC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Shangrong Fan, Profesor, Peking University Shenzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pkuszh-2020-02
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Vulvovaginal Candidiasis
Keywords: Recurrent Vulvovaginal Candidiasis; Lactobacillus; reproductive tract flora
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clotrimazole vaginal tablets (Active Comparator): Intensive treatment: clotrimazole vaginal tablets 500mg, every 72 hours, three consecutive times Consolidation treatment: clotrimazole vaginal tablets 500mg, once a week, 6 months
  Interventions: Drug: clotrimazole vaginal tablets
- Clotrimazole vaginal tablets+ Lactobacillus (Active Comparator): Intensive treatment: clotrimazole vaginal tablets 500mg, every 72 hours, three consecutive times + Lactobacillus Consolidation treatment: clotrimazole vaginal tablets 500mg, once a week, 6 months
  Interventions: Drug: Clotrimazole vaginal tablets+ Lactobacillus

INTERVENTIONS:
Drug: clotrimazole vaginal tablets — Intensive treatment: clotrimazole vaginal tablets 500mg, every 72 hours, three consecutive times Consolidation treatment: clotrimazole vaginal tablets 500mg, once a week, 6 months
  Other Names: clotrimazole vaginal tablets（Bayer）
  Arms: Clotrimazole vaginal tablets
Drug: Clotrimazole vaginal tablets+ Lactobacillus — Intensive treatment: clotrimazole vaginal tablets 500mg, every 72 hours, three consecutive times Consolidation treatment: clotrimazole vaginal tablets 500mg, once a week, 6 months Human Reproductive Tract Active Lactobacillus,4g,qd ,3months
  Other Names: Clotrimazole vaginal tablets+ Lactobacillus（Umeta-mimi）
  Arms: Clotrimazole vaginal tablets+ Lactobacillus

SUMMARY:
We are trying to determine if Clotrimazole vaginal tablets with oral Lactobacillus is better than Clotrimazole vaginal tablets in Preventing the Recurrence of vulvovaginalcandidiasis

DETAILED DESCRIPTION:
vulvovaginal candidiasis is common disease in women. Its refractory and high recurrence rate has always been a clinical problem. Some cases even recur several times a year, and those who recur more than four times a year are diagnosed as recurrent vaginal candidal infection Candidiasis, RVVC）。 The common clinical regimen for VVC is to strengthen and consolidate clotrimazole vaginal tablets for up to 25 weeks. However, long-term antibiotic treatment will lead to the decrease of vaginal microflora and the disappearance of inflammation and pathogenic bacteria, which will greatly increase the probability of repeated infection and become a barrier to clinical treatment. If probiotics are added in the treatment, the abundance of lactobacillus can be ensured while antibiotic treatment is carried out, the homeostasis of reproductive tract flora can be reestablished, the defense mechanism can be improved fundamentally, and the re invasion of pathogenic bacteria can be reduced, which will become a new treatment idea and method for radical cure of refractory RVVC.

We hypothesize that Clotrimazole vaginal tablets with oral Lactobacillus is better than Clotrimazole vaginal tablets in Preventing the Recurrence of vulvovaginalcandidiasis.

ELIGIBILITY:
Inclusion Criteria:

* Women be at least 18 years of age
* Have symptoms of vulva irritation and or abnormal discharge
* Meet the clinical criteria for RVVC
* Willing to participate in research

Exclusion Criteria:

1. Taking / injecting antibiotics in the past two weeks;
2. A woman who intends to be pregnant, pregnant or lactating;
3. Long term use of contraceptives and immunosuppressants;
4. Postmenopausal;
5. There was no same fixed sexual partner (RSP) before and after treatment
6. Patients with severe gastrointestinal diseases, including colorectal cancer, IBS, IBD, chronic or acute diarrhea, long-term constipation, etc., or receiving gastrointestinal surgery and abdominal surgery within one year, such as cholecystectomy;
7. Patients with severe heart, liver and kidney dysfunction, mental diseases, infectious diseases, tumors, severe anemia, and severe autoimmune diseases (such as rheumatoid arthritis, lupus erythematosus, etc.)

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The cure rate of RVVC, | 6 months
  The cure rate of RVVC,

SECONDARY OUTCOMES:
Recurrence of RVVC | 6 months
  Recurrence of RVVC

CONTACTS AND LOCATIONS:
Overall Officials: Shangrong Fan, M.D., Principal Investigator — Peking University Shenzhen Hospital
Locations (1):
- Dept Obstetrics and Gynecology, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No